CLINICAL TRIAL: NCT05259527
Title: Impact of Vitamin D Supplementation on Reported Rates of Taxane-Induced Neuropathy
Brief Title: Vitamin D Supplementation on Reported Rates of Taxane-Induced Neuropathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCC-21-18386; HM20023717 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic pain; Neuropathy; Vitamin-D
MeSH Terms: conditions — Neuralgia | interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vitamin D Replacement (Experimental): Participants will receive prescribed oral vitamin D2 to achieve a serum vitamin D level between 30 ng/mL to 50 ng/mL.
  Interventions: Drug: Ergocalciferol Capsules
- Standard of Care (Active Comparator): Participants will receive standard-of-care advice to take over the counter vitamin D.
  Interventions: Dietary Supplement: Cholecalciferol Capsules
- Observation Arm (No Intervention): Observation only

INTERVENTIONS:
Drug: Ergocalciferol Capsules — Vitamin D2 50,000IU by mouth once weekly for 8 weeks then once per month thereafter.
  Other Names: Vitamin D2
  Arms: Vitamin D Replacement
Dietary Supplement: Cholecalciferol Capsules — Vitamin D3 5,000IU by mouth daily
  Other Names: Over the Counter Vitamin D3
  Arms: Standard of Care

SUMMARY:
This is a two-arm randomized clinical trial in which 80 participants with Vitamin D deficiency and scheduled to begin taxane-based chemotherapy will be randomized to either: 1) prescribed vitamin D replacement or 2) standard of care.

DETAILED DESCRIPTION:
This is a two-arm randomized clinical trial in which 80 participants with Vitamin D deficiency and scheduled to begin taxane-based chemotherapy will be randomized to either: 1) prescribed vitamin D replacement or 2) standard of care (advised to take over the counter (OTC) vitamin D).

All participants will have blood drawn for serum vitamin D analysis at Weeks 4, 8, 12, and 24 in order to document Vitamin D levels and titrate vitamin D dose (if needed in the treatment arm). Participants in both arms will complete self-report measures of neuropathic pain at baseline, Week 12, and Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage I-III cancer of any type, OR diagnosis of stage IV cancer being treated with curative intent
* Receiving or scheduled to begin taxane-based chemotherapy at Virginia Commonwealth University (VCU) Health Massey Comprehensive Cancer Center
* Vitamin D serum level <20 ng/mL Note: study participants with Vitamin D serum level ≥20 ng/mL may be enrolled in the observational arm.

Exclusion Criteria:

* Pre-existing diagnosis of neuropathy
* Currently taking prescription Vitamin D (ergocalciferol)
* Inability to converse in English
* Pregnancy
* Chronic kidney disease (stage IV or greater)
* Known hyperparathyroidism
* Hypercalcemia: Calcium levels >10.5 mg/dL Note: study participants with calcium levels <10.5 mg/dL may be enrolled in the observational arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported neuropathic pain- sensory symptoms | 12 Weeks
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-CIPN (EORTC-QLQ-CIPN20) is a 20-item self-report questionnaire that includes a 9-item subscale assessing sensory symptoms of peripheral neuropathy. The questionnaire asks respondents to think about their past week and indicate to what extent they experienced symptoms of peripheral neuropathy: not at all; a little; quite a bit; or very much. The EORTC-QLQ-CIPN20 will be administered at baseline and at 12 weeks in order to assess change in scores over time.
Self-reported neuropathic pain- motor symptoms | 12 weeks
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-CIPN (EORTC-QLQ-CIPN20) is a 20-item self-report questionnaire that includes a 8-item subscale assessing motor symptoms of peripheral neuropathy. The questionnaire asks respondents to think about their past week and indicate to what extent they experienced symptoms of peripheral neuropathy: not at all; a little; quite a bit; or very much. The EORTC-QLQ-CIPN20 will be administered at baseline and at 12 weeks in order to assess change in scores over time.
Self-reported neuropathic pain- autonomic symptoms | 12 weeks
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-CIPN (EORTC-QLQ-CIPN20) is a 20-item self-report questionnaire that includes a 3-item subscale assessing autonomic symptoms of peripheral neuropathy. The questionnaire asks respondents to think about their past week and indicate to what extent they experienced symptoms of peripheral neuropathy: not at all; a little; quite a bit; or very much. The EORTC-QLQ-CIPN20 will be administered at baseline and at 12 weeks in order to assess change in scores over time.

SECONDARY OUTCOMES:
Self-reported neuropathic pain | 12 Weeks
  The number of participants with self reported neuropathic pain using the PROMIS Scale v. 2.0 - Neuropathic Pain Quality 5a. This 5-item questionnaire asks respondents to indicate the extent to which they experienced symptoms of peripheral neuropathy in the past week on a scale from 1 ("not at all") to 5 ("very much"). The PROMIS Scale v. 2.0 - Neuropathic Pain Quality 5a will be administered at baseline and at 12 weeks in order to assess change in scores over time.
Clinical diagnosis of peripheral neuropathy | 12 Weeks
  The number of participants with a clinical diagnosis of peripheral neuropathy. Chart review will be performed in order to determine whether an independent clinical diagnosis of peripheral neuropathy has been made for study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hong, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to make individual participant data (IPD) available to other researchers at this time.